CLINICAL TRIAL: NCT02864693
Title: Comparative Effectiveness of Microprocessor Controlled and Carbon Fiber Energy Storing and Returning Prosthetic Feet in Persons With Unilateral Transtibial Amputation
Brief Title: Comparative Effectiveness of Microprocessor Controlled and Carbon Fiber Prosthetic Feet in Transtibial Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ability Prosthetics and Orthotics, Inc. (Industry)
Responsible Party: Principal Investigator, Brian Kaluf BSE, CP, Clinical Outcome and Research Director, Ability Prosthetics and Orthotics, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FI-001
Record Dates: First submitted 2016-08-04; First posted 2016-08-12 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Amputation
Keywords: Microprocessor Controlled Ankle; Transtibial Amputee; Pacifica LP; Kinnex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Configuration A (Kinnex) (Active Comparator)
  Interventions: Device: Kinnex
- Configuration B (Pacifica LP) (Active Comparator)
  Interventions: Device: Pacifica LP

INTERVENTIONS:
Device: Kinnex — The Kinnex is a microprocessor controlled hydraulic ankle foot device (Freedom Innovations, Irvine, CA).
  Arms: Configuration A (Kinnex)
Device: Pacifica LP — The Pacifica LP is a carbon-fiber ankle foot device (Freedom Innovations, Irvine, CA)
  Arms: Configuration B (Pacifica LP)

SUMMARY:
The purpose of this research is to evaluate benefits of a microprocessor controlled prosthetic ankle-foot device compared to a non-microprocessor controlled or passive carbon fiber prosthetic ankle-foot device.

DETAILED DESCRIPTION:
Recent advancements in microprocessor controlled prosthetic ankle-foot systems have allowed additional functionality for the lower limb amputee, but research into the effectiveness of microprocessor controlled ankle-foot systems has been limited.

In this research study, differences in perceived mobility, functional capabilities and gait parameters between energy storing and returning and microprocessor controlled ankle-foot mechanisms will be identified where they exist. Also a comparison of the initial function with a new system compared to the function after a four week accommodation period will provide insight into the time it takes for the prosthesis user to experience a benefit from a microprocessor ankle-foot.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transtibial amputation
* Age 18-99 years old
* Body weight below 275 lbs
* Non-pregnant
* English speaking
* Current user of prosthesis for at least one year
* Wear time 8 hrs/day or more
* MFCL ≥ K-3
* Well-fitting and functioning prosthesis
* No use of ambulatory aide
* Able to tolerate testing protocol
* Able to walk on slopes
* Must, in the opinion of the investigator, be willing and able to complete all aspects of the study, adhere to the study visit schedule and comply with the assessments

Exclusion Criteria:

* Amputation level other than unilateral transtibial
* Age <18 or >99 years old
* Body weight above 275 lbs
* Pregnant
* Non-English speaking
* Not current user of prosthesis
* Less than one year use of prosthesis
* Wear time less than 8 hr/day
* MFCL <K3
* Poor fitting and functioning prosthesis
* Indicating that the socket fit is painful, or unacceptable
* Use of ambulatory aide
* Unable to tolerate testing protocol
* Unable to walk on slopes
* Presence or history of any condition that, in the view of the investigator, places the participant at high risk of poor treatment compliance or of not completing the study
* Any neurologic impairments known to cause gait and/or balance dysfunction

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Amputee Mobility Predictor with Prosthesis (AMPPRO) | Collection at baseline
  The AMPPRO is a functional test consisting of 21 tasks that are similar to everyday function to test balance, strength and walking ability
L-Functional Test (L-Test) Baseline | Collection at baseline
  The L-test is a timed functional test that involves standing from a chair, walking 3 meters, turning around and sitting back into the chair.
5 times Sit-to-Stand (5 times STS) Baseline | Collection at baseline
  The 5 times STS is a timed functional test that measures how long it takes to stand and sit five times in a row from a chair.
6 minute Timed Walk Test (6m TWT) Baseline | Collection at baseline
  The 6m TWT involves walking as far as possible along a straight path between two cones in under 6 minutes.
Physiological Cost Index (PCI) Baseline | Collection at baseline
  The PCI is calculated by subtracting resting heart rate from active heart rate following a walking test, and dividing the difference by the walking speed.
Hill Assessment Index (HAI) Baseline | Collection at baseline
  The HAI is a functional test that measures quality of walking up and down a sloped ramp.
2 Dimensional Video Motion Analysis (2D Video Analysis) Baseline | Collection at baseline
  2D Video Analysis will be used to measure knee and ankle angles at mid-stance of gait while walking up and down the sloped ramp and also while standing still on level ground.
L-Functional Test (L-Test) after 4 weeks | Collection after 4 weeks
  The L-test is a timed functional test that involves standing from a chair, walking 3 meters, turning around and sitting back into the chair.
5 times Sit-to-Stand (5 times STS) after 4 weeks | Collection after 4 weeks
  The 5 times STS is a timed functional test that measures how long it takes to stand and sit five times in a row from a chair.
6 minute Timed Walk Test (6m TWT) after 4 weeks | Collection after 4 weeks
  The 6m TWT involves walking as far as possible along a straight path between two cones in under 6 minutes.
Physiological Cost Index (PCI) after 4 weeks | Collection after 4 weeks
  The PCI is calculated by subtracting resting heart rate from active heart rate following a walking test, and dividing the difference by the walking speed.
Hill Assessment Index (HAI) after 4 weeks | Collection after 4 weeks
  The HAI is a functional test that measures quality of walking up and down a sloped ramp.
2 Dimensional Video Motion Analysis (2D Video Analysis) after 4 weeks | Collection after 4 weeks
  2D Video Analysis will be used to measure knee and ankle angles at mid-stance of gait while walking up and down the sloped ramp and also while standing still on level ground.

SECONDARY OUTCOMES:
Orthotic Prosthetic User Survey (OPUS) | Collection after 4 weeks
  The OPUS is a self-reported questionnaire that asks about satisfaction with device
Prosthesis Evaluation Questionnaire - Mobility Subscale (PEQ-MS) | Collection after 4 weeks
  The PEQ-MS is a self-reported questionnaire that measures perceived difficulty ambulating on a variety of environmental barriers
Prosthesis Limb User Survey of Mobility (PLUS-M) | Collection after 4 weeks
  The PLUS-M is a self-reported questionnaire that measures perceived mobility with a prosthesis in different environments.
Activities-Specific Balance Confidence Scale (ABC) | Collection after 4 weeks
  The ABC is a self-reported questionnaire that measures confidence in balance while performing various activities in different environments.
Socket Comfort Score (SCS) | Collection at baseline and after 4 weeks
  The SCS is a self-reported questionnaire that asks the participant to rate their current socket comfort from 0-10, with 10 points representing the most comfortable socket they can imagine.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Ability Prosthetics and Orthotics, Inc. - Hagerstown, MD, Hagerstown, Maryland
  - Ability Prosthetics and Orthotics, Inc. - Charlotte, NC, Charlotte, North Carolina
  - Ability Prosthetics and Orthotics, Inc. - York, PA, York, Pennsylvania

IPD SHARING:
Plan to Share IPD: No